CLINICAL TRIAL: NCT06273150
Title: Dentatorubral-pallidoluysian Atrophy Natural History and Biomarkers Study
Acronym: DRPLA NHBS
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 142048
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Dentatorubral-Pallidoluysian Atrophy
Keywords: Dentatorubral-Pallidoluysian Atrophy; Ataxia; Epilepsy; Chorea
MeSH Terms: conditions — Myoclonic Epilepsies, Progressive; Ataxia; Epilepsy; Chorea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, CSF, saliva, urine, faeces, and fibroblasts
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DRPLA-mutation carrier: Subjects with a positive genetic test for a pathological expansion in the ATN1 gene.
  Interventions: Other: Positive genetic test for pathological expansion in ATN1
- Volunteer control: Subjects without neurological conditions (other than primary headache disorders), without a family history of DRPLA or a previous negative genetic test for pathological expansions in the ATN1 gene.
  Interventions: Other: Positive genetic test for pathological expansion in ATN1

INTERVENTIONS:
Other: Positive genetic test for pathological expansion in ATN1 — Positive genetic test for pathological expansion in ATN1

SUMMARY:
DRPLA Natural History and Biomarkers Study (DRPLA NHBS) is a prospective observational study that will lay the foundation for clinical trials in DRPLA. The aims of this project are:

* To characterize the natural history of DRPLA in both juvenile- and adult-onset patients and study different modalities of biomarkers in this condition.
* To identify genetic factors and biomarkers that could predict disease progression.
* To provide a platform to support the design and conduct of clinical trials.

This study has three arms:

1. Adult Participants: this arm of the study will require participants to be 16 years old or over to participate.
2. Pediatric Participants: this arm of the study will require participants to be under 16 years old to participate.
3. Remote Participants: patients that cannot or do not wish to travel to one of the study sites can participate in this arm of the study, irrespective of their age.

Participants will have an annual visit for three years (baseline visit and two follow-up visits, three visits in total). Subjects who complete the whole protocol will be assessed on two consecutive days to reduce patient burden.

This project will allow for a better understanding of DRPLA and its course, and therefore allow for future clinical trials on this condition to be more precisely and effectively conducted.

ELIGIBILITY:
Inclusion criteria for the Adult Protocol:

1. DRPLA adult participants must be 16 years old or over at the time of enrollment, to participate.
2. DRPLA adult participants must have a genetic diagnosis of DRPLA and CAG repeat expansion >35.
3. Patient is able to read, understand, and provide written informed consent (signed and dated). If the patient is under the age of 18 or is unable to provide consent, the patient must have a parent or caregiver capable of providing informed consent (signed and dated) and able to attend all scheduled study visits, and provide feedback regarding the participant's symptoms and performance as described in the protocol.
4. Adult pre-symptomatic subjects must have a positive genetic test for the DRPLA expansion without symptoms compatible with the disease, and be 16 years old or over at the time of enrollment.
5. Adult Family/Community control participants must be 16 years old or over at the time of enrollment to participate. Blood-relatives must not have a genetic diagnosis of DRPLA or their genetic status is unknown.

Exclusion criteria for the Adult Protocol:

1. Individuals with an ataxia condition other than DRPLA.
2. Failure to sign the consent form will result in study exclusion.
3. Has any condition or circumstance that, in the opinion of the Investigator, makes the participant unsuitable for enrolment. These may include medical conditions which might affect the measurement of biomarkers.
4. Participants will be excluded from the lumbar puncture, and skin biopsy procedures if they have a history of severe allergic or anaphylactic reactions or other adverse reactions to local anesthetics used in the study.
5. For family/community controls: those individuals with neurological conditions (other than primary headache disorders) will be excluded.

Inclusion Criteria for the Pediatric Protocol:

a. DRPLA pediatric participants must be under 16 years old at the time of enrollment, to participate.

f. DRPLA pediatric participants must have a genetic diagnosis of DRPLA and CAG repeat expansion >35.

g. If the patient is under the age of 18 or is unable to provide consent, the patient must have a parent or caregiver capable of providing informed consent (signed and dated) and able to attend all scheduled study visits, and provide feedback regarding the participant's symptoms and performance as described in the protocol.

h. Pediatric Family/Community control participants must be under 16 years old at the time of enrollment to participate. Blood-relatives must not have a genetic diagnosis of DRPLA or their genetic status is unknown.

Exclusion Criteria for the Pediatric Protocol:

f. Individuals with an ataxia condition other than DRPLA. g. Failure to sign the consent form will result in study exclusion. h. Has any condition or circumstance that, in the opinion of the Investigator, makes the participant unsuitable for enrolment. These may include medical conditions which might affect the measurement of biomarkers.

i. Participants will be excluded from the lumbar puncture, and skin biopsy procedures if they have a history of severe allergic or anaphylactic reactions or other adverse reactions to local anesthetics used in the study.

j. For family/community controls: those individuals with neurological conditions (other than primary headache disorders) will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community and/or clinical sample
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Scale for the assessment and rating of ataxia (SARA) | 3 years
  Progression of ataxia is measured using a validated ataxia scale, SARA. Scores range from 0 (no ataxia) to 40 (most severe ataxia).
Brain atrophy | 3 years
  Brain MRI is used to measure atrophy. Atrophy is expected to be observed in DRPLA patients, and in particular in the brainstem, superior cerebellar peduncle, cerebellum and thalamus.
Neurofilament plasma concentration (NfL) | 3 years
  Blood and CSF samples will be measured for NfL, a brain-derived protein.

SECONDARY OUTCOMES:
Inventory of non-ataxia signs (INAS) | 3 years
  The occurrence of accompanying non-ataxia symptoms is assessed using INAS.
Upper limb function test AIM-S | 3 years
  Hand dexterity and upper limb function is assessed using the AIM-S spoon test.
Redenlab DRPLA specific speech battery | 3 years
  Speech is assessed using the Redenlab software speech battery.
Clinical Assessment of Dysphagia in Neurodegeneration (CADN) | 3 years
  Dysphagia is assessed using the CADN, an assessment of swallowing in neurodegenerative disease.
Tau plasma concentration | 3 years
  Blood and CSF samples will be measured for Tau, a brain-derived protein.
Glial fibrillary acidic protein (GFAP) concentration | 3 years
  Blood and CSF samples will be measured for GFAP, a brain-derived protein.
Ubiquitin carboxyterminal hydrolase L1 (UCH-L1) concentration | 3 years
  Blood and CSF samples will be measured for UCH-L1, a brain-derived protein.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Giunti, Principal Investigator — University College, London
Locations (3):
- United States (2):
  - NYU Grossman School of Medicine, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be decided upon publication of study results and agreements with other researchers.